CLINICAL TRIAL: NCT03414398
Title: Assessing Cirrhosis Quality of Care While Accounting for Cost: Is the Patient and/or Caregiver Perspective Associated With Outcomes or Quality Metrics, and What is the Cost of Implementing and Measuring Quality Metrics
Brief Title: Assessing Cirrhosis Quality of Care While Accounting for Cost
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: New York Presbyterian Hospital (Other)
Responsible Party: Principal Investigator, Nicole T Shen, Principal Investigator, New York Presbyterian Hospital
Other Study IDs: 1710018603
Record Dates: First submitted 2017-12-26; First posted 2018-01-30 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental: Qualitative interview

SUMMARY:
The objective of this study is to determine what influences the patient and caregiver perception of care, and if this perception associates with the percentage of and what quality metrics are being met and outcomes. The investigators also plan to capture the cost of providing quality metrics and the cost of monitoring adherence to quality metrics.

DETAILED DESCRIPTION:
This study will be conducted using mixed-methods. The qualitative part will consist of in person, 1:1, open ended in depth interviews using a standard interview guide with probes. The quantitative part will document subjects meeting or not meeting the quality metrics supported by strong evidence, clinical outcomes, and medical bills.

ELIGIBILITY:
Inclusion Criteria:

* primary liver cirrhosis
* receiving care at the study cite
* no evidence of hepatic encephalopathy if the subject is providing consent

Exclusion Criteria:

* no documentation of cirrhosis
* unable to confirm diagnosis of cirrhosis by imaging or pathology

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Cirrhosis, aged 18-80.
Sampling Method: Non-Probability Sample
Enrollment: 273 (Estimated)
Dates: Start 2017-12-26 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Participant perceptions of care | 2 years
  Qualitative interview performed where the participant describes their experience of the quality of care they have received.
Relationship of perceptions of quality of care to recent hospitalizations | 2 years
  Assess associations of qualitative themes that emerge from the qualitative interview with hospitalization frequency
Relationship of perceptions of quality of care to portal hypertension quality metric adherence | 2 years
  Assess associations of qualitative themes that emerge from the qualitative interview with physician meeting of portal hypertension quality metric (i.e., physician follows the recommended management (yes/no)).

SECONDARY OUTCOMES:
Assess if portal hypertension quality metric adherence equates to less hospitalizations | 2 years
  To see if there is an association of portal hypertension quality metric adherence (i.e. physician follows the recommended management of portal hypertension (yes/no)) to frequency of hospitalizations.
Association of quality metric adherence with survival | 2 years
  We will explore adherence with proposed portal hypertension quality metric (physician follows the management (yes/no)) to see if there is an association with survival. The quality metric will be identified as either being met or not met, and survival will also be identified as having occurred or not.

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Brown, MD, MPH, Principal Investigator — New York Presbyterian Hospital - Weill Cornell
Locations (1):
- New York Presbyterian Hospital - Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No